CLINICAL TRIAL: NCT06504498
Title: The Effectiveness of Orthodontic Treatment With Clear Aligners in Different Thicknesses
Brief Title: Effectiveness of Clear Aligners in Different Thicknesses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Saniye Merve CENGIZ, Assistant Professor, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MEÜ-SCENGİZ-01
Record Dates: First submitted 2024-06-28; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Angle's Class I Malocclusion; Crowding, Tooth
Keywords: Clear aligner thickness; Orthodontic tooth movement; Pain
MeSH Terms: conditions — Malocclusion, Angle Class I; Malocclusion; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.5 mm-thick Duran® clear aligners (Active Comparator): 0.5 mm-thick clear aligners (Duran®; Scheu-Dental GmBH, Iserlohn, Germany).
  Interventions: Device: 0.5 mm-thick Duran® clear aligner
- 0.75 mm-thick Duran® clear aligners (Experimental): 0.75 mm-thick clear aligners (Duran®; Scheu-Dental GmBH, Iserlohn, Germany).
  Interventions: Device: 0.75 mm-thick Duran® clear aligner

INTERVENTIONS:
Device: 0.5 mm-thick Duran® clear aligner — 0.5 mm-thick clear aligner was used for orthodontic treatment.
  Arms: 0.5 mm-thick Duran® clear aligners
Device: 0.75 mm-thick Duran® clear aligner — 0.75 mm-thick clear aligner was used for orthodontic treatment.
  Arms: 0.75 mm-thick Duran® clear aligners

SUMMARY:
This study aimed to evaluate the effectiveness, pain, and satisfaction levels between patients treated with different thicknesses of clear aligners among Class I maxillary mild crowding cases. Two types of clear aligners with thicknesses of 0.5 and 0.75 mm were used. The null hypotheses were as follows: There is no clinical difference in effectiveness, pain, and satisfaction levels between different thickness of clear aligners. The alternate hypotheses were as follows: The thicker the clear aligner, the greater orthodontic force applied to tooth which affects the amount of orthodontic tooth movement, pain, and satisfaction levels of patients. The primary aim was to evaluate pre- and post-treatment changes in amount of orthodontic tooth movement. Maxillary cephalometric parameters were measured on lateral cephalograms and maxillary dental parameters were measured using OrthoAnalyzer, and compared before and after treatment. Visual Analogue Scale and Patient Satisfaction Evaluation Form were used in order to assess the pain and satisfaction levels of patients. Pain and satisfaction levels were measured before the aligner insertion (T0), at the 4th hour (T1), 2nd day (T2), 1st week (T3), 1st month (T4) and at the end of the treatment (T5).

DETAILED DESCRIPTION:
The sample size was computed to detect difference in the amount of orthodontic tooth movement between groups (G*Power, University of Dusseldorf, Germany). The calculated sample size was 14 for each group, similar to the previously published study (effect size = 0.8, α = 0.05, and 1 - β = 0.80). Lateral cephalograms were taken for all patients using the X-ray device (PM 2002 EC Proline; Planmeca OY, Helsinki, Finland) in the Department of Oral and Maxillofacial Radiology. Patients who satisfied the inclusion criteria were enrolled in this study and they were randomly separated into 2 groups (Group 1 and Group 2) based on the aligner thickness, each consisted of 14 patients. Patients in Group 1 were treated with 0.5 mm-thick clear aligners, patients in Group 2 were treated with 0.75 mm-thick clear aligners. The Little's Irregularity Index were calculated using OrthoAnalyzer software (3Shape, Copenhagen, Denmark) to standardize the amount of maxillary anterior crowding at the beginning of the treatment. Initial records were taken at the beginning of the treatment using an intraoral scanner (Trios 3®, 3Shape, Copenhagen, Denmark). Scanned data has been converted to standard tessellation language (STL) files and these files have been modified to create virtual setups for orthodontic tooth movement using OrthoAnalyzer software. Virtual setups were imported into a slicing software for model preparation before printing. A stereolithographic (SLA) 3D printer and liquid photopolymer were used to print resin models. These models were used as mould for thermoforming of the aligners using a vacuum-thermoforming machine (Model No: 202, Keystone Industries, Myerstown, USA). All aligners were manually cut with straight trim lines at gingival zenith to provide better comfort for the patients. Attachments were placed according to the software and interproximal reductions were performed by the same operator (SMC). Patients were followed at 2nd day (T2), 1st week (T3), 1st month (T4) and at the end of the treatment (T5). Pre- (T0) and post-treatment (T5) digital models, lateral cephalometric radiographs were compared. Pain and satisfaction levels of patients were assessed using Visual Analogue Scale and Patient Satisfaction Evaluation Form.

ELIGIBILITY:
Inclusion Criteria:

1. Angle Class I malocclusion without skeletal discrepancy,
2. Patients older than 18 years old with a full permanent dentition without supernumerary missing or impacted teeth except for 3rd molars,
3. Non-extraction cases with mild crowding in maxillary arch (2-5 mm),
4. Good oral health without periodontal disease or caries,
5. No previous orthodontic treatment,
6. Not taking pain medications.

Exclusion Criteria:

1. History of previous orthodontic or interceptive treatment,
2. Extraction cases with crowding of > 5 mm,
3. Presence of anterior or posterior openbite or crossbite,
4. Unwilling to be treated with clear aligners,
5. Presence of supernumerary, missing or impacted teeth (other than third molars),
6. Presence of any local/systemic problems or trauma, which may affect the pain level.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Radiographic tooth movement | At 6th months
  Changes in the amount of maxillary cephalometric parameters using lateral cephalometric radiographs after 6 months.
Orthodontic tooth movement | At 6th months
  Changes in intercanine, interpremolar, intermolar arch expansions and dental arch perimeter (maxillary dental parameters) using OrthoAnalyzer® software after 6 months.

SECONDARY OUTCOMES:
Patients' pain level | At the 4th hours, 2nd days, 1st week, 1st month, and 6th months
  Changes in patients' pain level using a 10-cm VAS using ''no pain'' and ''severe pain'' as anchor descriptions at the 4th hours, 2nd days, 1st week, 1st month, and 6th months.
Patients' satisfaction level | At the 4th hours, 2nd days, 1st week, 1st month, and 6th months
  Changes in patients' satisfaction level using ''Patient Satisfaction Evaluation Form 1'' at the 4th hours, 2nd days, 1st week, 1st month; and using ''Patient Satisfaction Evaluation Form 2'' at the 6th months.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Göymen, Assoc Prof, Study Director — Study Director
Locations (1):
- Mersin University Faculty of Dentistry Department of Orthodontics, Mersin, Turkey (Türkiye)

REFERENCES:
- [Result] Sachdev S, Tantidhnazet S, Saengfai NN. Accuracy of Tooth Movement with In-House Clear Aligners. J World Fed Orthod. 2021 Dec;10(4):177-182. doi: 10.1016/j.ejwf.2021.08.003. Epub 2021 Oct 5. PMID 34625386
- [Result] Ho CT, Huang YT, Chao CW, Huang TH, Kao CT. Effects of different aligner materials and attachments on orthodontic behavior. J Dent Sci. 2021 Jul;16(3):1001-1009. doi: 10.1016/j.jds.2021.01.011. Epub 2021 Feb 12. PMID 34141116
- [Derived] Cengiz SM, Goymen M. The effectiveness of orthodontic treatment with clear aligners in different thicknesses. Sci Rep. 2025 Feb 1;15(1):3958. doi: 10.1038/s41598-025-86345-9. PMID 39893227